CLINICAL TRIAL: NCT00141206
Title: A Twelve-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study With Follow-up Evaluating the Safety and Efficacy of Varenicline Tartrate ( CP-526,555) in Comparison to Zyban for Smoking Cessation
Brief Title: A Twelve-Week Study of Varenicline for Safety and Efficacy in Comparison With Placebo and Zyban for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051028
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline (CP-526,555)

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of varenicline given for a twelve week treatment period in comparison with placebo and Zyban for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects who have used bupropion (Zyban, or Wellbutrin) previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005
Dates: Start 2003-05; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
4 week Continuous Quit Rate ( 4 week CQR ) for weeks 9 -12

SECONDARY OUTCOMES:
Continuous abstinence Weeks 9-52
Long-term Quit Rate Week 52
Continuous abstinence Weeks 9 -24
7-day Point Prevalence Abstinence Weeks 12, 24, and 52
4-week Point Prevalence Abstinence at Week 52
Minnesota Nicotine Withdrawal Scale
Brief Questionnaire of Smoking Urges
Smoking Effects Inventory
Change from baseline in bodyweight

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hays JT, Croghan IT, Baker CL, Cappelleri JC, Bushmakin AG. Changes in health-related quality of life with smoking cessation treatment. Eur J Public Health. 2012 Apr;22(2):224-9. doi: 10.1093/eurpub/ckq137. Epub 2010 Sep 30. PMID 20884658
- [Derived] Gonzales D, Jorenby DE, Brandon TH, Arteaga C, Lee TC. Immediate versus delayed quitting and rates of relapse among smokers treated successfully with varenicline, bupropion SR or placebo. Addiction. 2010 Nov;105(11):2002-13. doi: 10.1111/j.1360-0443.2010.03058.x. Epub 2010 Sep 1. PMID 20819082
- [Derived] Hays JT, Leischow SJ, Lawrence D, Lee TC. Adherence to treatment for tobacco dependence: association with smoking abstinence and predictors of adherence. Nicotine Tob Res. 2010 Jun;12(6):574-81. doi: 10.1093/ntr/ntq047. Epub 2010 May 10. PMID 20457644
- [Derived] Nides M, Glover ED, Reus VI, Christen AG, Make BJ, Billing CB Jr, Williams KE. Varenicline versus bupropion SR or placebo for smoking cessation: a pooled analysis. Am J Health Behav. 2008 Nov-Dec;32(6):664-75. doi: 10.5555/ajhb.2008.32.6.664. PMID 18442345
- [Derived] West R, Baker CL, Cappelleri JC, Bushmakin AG. Effect of varenicline and bupropion SR on craving, nicotine withdrawal symptoms, and rewarding effects of smoking during a quit attempt. Psychopharmacology (Berl). 2008 Apr;197(3):371-7. doi: 10.1007/s00213-007-1041-3. Epub 2007 Dec 15. PMID 18084743
- [Derived] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051028&StudyName=A+Twelve%2DWeek+Study+of+Varenicline+for+Safety+and+Efficacy+in+Comparison+with+Placebo+and+Zyban+for+Smoking+Cessation